CLINICAL TRIAL: NCT06653985
Title: Intra-articular Corticosteroid With Hyaluronic Acid Plus Physiotherapy for Hip Pathologies (NON-OP HIP) - a Randomized Controlled Trial
Brief Title: Intra-articular Corticosteroid With Hyaluronic Acid Plus Physiotherapy for Hip Pathologies (NON-OP HIP)
Acronym: NON-OP HIP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ArthroBiologix Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: nonophip
Record Dates: First submitted 2024-10-09; First posted 2024-10-23 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Osteoarthritis; Femoroacetabular Impingement Syndrome; Labrum Injury of the Hip Joint
Keywords: Hip; Osteoarthritis; Femoroacetabular impingement; Labral tear; Hyaluronic acid; Corticosteroid; Physical Therapy; Physiotherapy
MeSH Terms: conditions — Osteoarthritis; Femoracetabular Impingement | interventions — Adrenal Cortex Hormones; Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Hyaluronic and corticosteroid injection with physical therapy (Experimental): Patients will receive an ultrasound-guided injection consisting of 3 ml hyaluronic acid (Durolane™) mixed with 40 mg triamcinolone (Kenalog™) into their hip joint. Patients will also receive an 8-week physiotherapy protocol, consisting of 8 visits. The protocol will consist of 1 visit per week.
  Interventions: Drug: Hyaluronic and corticosteroid injection; Other: Physical Therapy
- Hyaluronic and corticosteroid injection (Active Comparator): Patients will receive an ultrasound-guided injection consisting of 3 ml hyaluronic acid (Durolane™) mixed with 40 mg triamcinolone (Kenalog™) into their hip joint.
  Interventions: Drug: Hyaluronic and corticosteroid injection

INTERVENTIONS:
Drug: Hyaluronic and corticosteroid injection — Patients will receive an ultrasound-guided injection consisting of 3 ml hyaluronic acid (Durolane™) mixed with 40 mg triamcinolone (Kenalog™) into their hip joint.
Other: Physical Therapy — Patients will receive an 8-week physiotherapy protocol, consisting of 8 visits. The protocol will consist of 1 visit per week.
  Arms: Hyaluronic and corticosteroid injection with physical therapy

SUMMARY:
Hip pathologies that cause pain and functional limitations are common in the general population. These can include femoroacetabular impingement (FAI), labral tears and mild osteoarthritis (OA) among others. While more severe and symptomatic cases may require surgical intervention, the treatment of mild-to-moderate cases is often treated without surgery to relieve pain, improve function, and delay surgical intervention.

Non-operative treatments of hip pathologies consist of a multitude of options. A common non-operative intervention includes intra-articular injections, including corticosteroids and hyaluronic acid. Evidence has demonstrated that corticosteroids have fast acting effects which tend to diminish within a few months, while hyaluronic acid has a delayed time of onset and demonstrates clinical benefit for a longer period of time. Studies have evaluated combinations of corticosteroid and hyaluronic acid, hoping to take advantage of the fast-acting relief of corticosteroid and the longer lasting benefits of corticosteroid.

Physiotherapy is also a frequent non-operative intervention used to relieve pain and increase function in patients with hip pathologies. While many studies have looked at intra-articular injections and physiotherapy as independent non-operative possibilities for hip conditions, the combined effect of these two have not received much evaluation. The purpose of this study is to evaluate the effect of physiotherapy in conjunction with a combined corticosteroid and hyaluronic acid intraarticular injection on patient outcomes when compared to a corticosteroid and hyaluronic acid intraarticular injection alone.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 40-60 years old.
2. Patients with mild hip arthritis (Kellgren-Lawrence grade 2 or lower) with or without a labral tear and/or femoroacetabular impingement and/or mild hip dysplasia.
3. Patients who demonstrate more than 50% reduction in hip pain following a diagnostic injection (ultrasound guided intra-articular anaesthetic only).
4. Able to subsidize private physiotherapy services.
5. Able to provide informed consent.

Exclusion Criteria:

1. Active infection
2. Osteonecrosis of the hip, moderate to severe arthritis (Kellgren-Lawrence grade 3 or higher), or moderate-to-severe hip dysplasia
3. Previous hip fracture, pelvic fracture, or lower limb fracture,
4. Previous surgery to the pelvis, hip or lower limb
5. Hypermobility disorder or connective tissue disease (e.g. Ehler's-Danlos syndrome, Marfan's syndrome etc.)
6. Patients with chronic low back pain and/or sciatica
7. Patients who received an intra-articular steroid hip injection within 3 months
8. Patients who have previously received a hyaluronic acid injection
9. Injuries sustained in a motor vehicle collision.
10. Injuries sustained in the workplace and have a worker's compensation claim.
11. Injuries resulting in a medico-legal dispute.
12. Patients who are pregnant of planning to become pregnant
13. Currently enrolled in a study that does not permit co-enrollment
14. Unable to obtain informed consent
15. Unable to comply with the study protocol
16. Contraindication to corticosteroid or hyaluronic acid injection
17. Prior enrollment in the study.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | 6 months post-injection
  NPRS is scored by asking the patient to circle the number between 0 and 10 that fits best to their pain intensity. Zero represents "no pain" whereas the upper limit of 10 represents "worst possible pain". The patient score is determined as a score out of 10 based on where they indicate their pain falls by selecting a number between 0 and 10 which most accurately represents their pain.

SECONDARY OUTCOMES:
International Hip Outcome Tool 12 item (iHOT-12) | 6 months post-injection
  The tool consists of 12 VAS questions evaluating 4 areas: symptoms and functional limitations, sports and recreational activities, job-related concerns, and social, emotional, and lifestyle concerns. The patient score is determined by averaging the score of the 12 items in the iHOT-12 and is presented on a scale of 0-100, with 0 representing the worst possible function and 100 representing the best possible function.
EuroQol-5D-5L (EQ-5D) | 6 months post-injection
  A quality-of-life measurement instrument that provides a score based on 5 dimensions of quality of life: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. This brief questionnaire is self-reported by the patient and determines a quality of life score between 0 and 1, where 1 represents perfect health and 0 represents death.
Medication Use | 6 months post-injection
  Patient medication use, including types (analgesics, NSAIDs, opioids) will be asked at baseline. Patient will then be asked at 3- and 6- months if they are currently using pain medication, and if so whether their use has decreased, stayed the same, or increased.
Adverse Events | 6 months post-injection
  Adverse events experienced over the course of the study will be documented.

CONTACTS AND LOCATIONS:
Locations (1):
- ArthroBiologix, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No